CLINICAL TRIAL: NCT04532710
Title: Clinical Evaluation of Two Different Dosage Groups of Tacrosolv Eye Drops in a Placebo Controlled Crossover Design to Evaluate Safety and Efficacy in Patients Suffering From Grass Pollen Induced Allergic Rhinoconjunctivitis in the Vienna Challenge Chamber.
Brief Title: Therapeutic Effect of Tacrosolv in Patients With Allergic Rhinoconjunctivitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinomed Biotech AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCS_19_02; 2019-002847-62 (EudraCT Number)
Record Dates: First submitted 2020-08-21; First posted 2020-08-31 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Allergic Conjunctivitis; Allergic Rhinitis
Keywords: Conjunctivitis; Allergic rhinoconjunctivitis; Tacrolimus; Allergen exposure chamber; Total Ocular Symptom Score; Onset of action; Tacrosolv; Ocular redness; Vienna Challenge Chamber
MeSH Terms: conditions — Conjunctivitis, Allergic; Rhinitis, Allergic; Conjunctivitis | interventions — Ophthalmic Solutions; Solutions

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, double-blind, single site trial in a validated allergen exposure chamber setting using grass pollen induced rhinoconjunctivitis.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo low dose (Placebo Comparator): Application of 2 placebo eye drops once daily for 8 days.
  Interventions: Drug: Eye Drops, Solution in Single-Dose Container
- Tacrosolv low dose (Active Comparator): Application of 1 Tacrosolv eye drop once daily for 8 days.
  Interventions: Drug: Eye Drops, Solution in Single-Dose Container
- Placebo high dose (Placebo Comparator): Application of 1 placebo eye drop once daily for 8 days.
  Interventions: Drug: Eye Drops, Solution in Single-Dose Container
- Tacrosolv high dose (Active Comparator): Application of 2 Tacrosolv eye drops once daily for 8 days.
  Interventions: Drug: Eye Drops, Solution in Single-Dose Container

INTERVENTIONS:
Drug: Eye Drops, Solution in Single-Dose Container — Application of eye drops

SUMMARY:
Allergic conjunctivitis is one of the most common comorbidities of allergic diseases, especially of allergic rhinitis.

Rhinoconjunctivitis is an allergic condition of the nasal mucosa and the eyes. Conjunctivitis is triggered by hypersensitivity to certain pollens and other airborne allergens and causes several symptoms such as reddened eyes, itchy eyes and can cause watery eyes and a scratchy feeling in the eye. Tacrolimus is a well-known immunosuppressiv active substance which is hardly soluble in water. Within Tacrosolv, Tacrolimus is completely dissolves in aqueous solution. The effectiveness of Tacrosolv will be tested for treatment of allergic conjunctivitis. Allergic subjects will be treated with aqueous formulation of tacrolimus 'Tacrosolv 50 micrograms per milliliter, eye drops' for 8 days. On day 1 and day 8 allergic patients will be challenged with grass pollen for a period of 4 hours and subjective allergic symptoms will be assessed.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, crossover, double-blind, single site trial in adult subjects (18-65 years of age) who have demonstrated grass specific Immunglobulin E (IgE) reactivity and have a history of grass pollen induced rhinoconjunctivitis with or without controlled asthma. The crossover design will ensure that individual subjects will receive either one drop Tacrosolv compared to two drops placebo or 2 drops Tacrosolv compared to 1 drop placebo.

The primary objective of the trial is to demonstrate the safety and efficacy of two doses of Tacrosolv on day 8 of treatment. To assure full blinding, two study populations are treated in a crossover design against placebo.

The evaluation will be based on the assessment of ocular symptoms during grass pollen challenge performed in the Vienna Challenge Chamber (environmental exposure chamber).

Secondary objective of the trial is to evaluate the onset of action of either dose of Tacrosolv on day one of treatment as well as efficacy differences between low dose and high dose treatment on day eight.

Visit 1 - Screening:

At least one week prior to first treatment block, subjects will be screened for appropriate allergic response during a grass pollen challenge chamber session. A total ocular symptom score (TOSS) of at least 4 points out of 12 within the first two hours in the grass pollen challenge chamber is required to be included into the study.

Visit 2 - Inclusion:

In addition to the screening provocation the medical and allergic history, safety lab as well as retrieving inclusion and exclusion criteria will be assessed via anamnesis. Furthermore, all safety assessments will be conducted.

Note: Visit 1 and visit 2 could be done on the same day!

Visit 3 & 5: Day1 of the respective treatment period

Eligible subjects will be randomly assigned to one of the four treatment arms (fully blinded) in the order of their screening numbers assigned at visit 1.

Subjects will attend the study site about two hours ahead of the start of allergen provocation. After positive completion of all study relevant assessments, baseline values for symptom scores will be assessed approximately 45 minutes before entering the grass pollen challenge chamber. Subjects will receive their first treatment 30 minutes before entering the challenge chamber. During the 4 hours grass pollen challenge subjective and objective assessments will be recorded.

The subjective ocular symptom score, as well as the other symptom scores, will be recorded every fifteen minutes during a 4-hour allergen exposure challenge. Before and after provocation session several ocular assessments will be performed.

After the allergen challenge, subjects will receive study medication for the home treatment phase (days 2 to 7) and continue treatment into each conjunctival sac once a day (in the morning) until day 7.

Visit 4 & 6: Day8 of respective treatment period

On day 8 of their respective treatment block, subjects will attend the study site about two hours before provocation starts. Before receiving their last treatment dose, baseline symptom scores will be assessed. Subjects will take their last treatment dosage approximately half an hour before entering the challenge chamber for a 4-hour allergen exposure challenge. Subjective symptom scores will be recorded every fifteen minutes. Slit lamp biomicroscopy including all other ocular assessments as mentioned above will be performed before and after the provocation session.

Between the respective study treatments, a wash-out period of at least 13 days must be adhered to allowing complete dissipation of the previous treatment.

After the wash-out period, subjects change to their respective next treatment block.

During the entire trial, subjects will be asked to monitor for adverse events (AEs), and they will record the use of concomitant medications on the provided form. Female subjects of child-bearing potential will complete a urine pregnancy test during screening and on D1 of each treatment period.

Following parameters will be assessed:

* Subjective symptom score (nasal, ocular, respiratory) during the grass pollen challenge lasting for 4 hours - every 15 minutes
* Active anterior rhinomanometry (AAR) - every 60 minutes
* Lung function tests using regular spirometry for FEV1 and FVC - every 60 minutes
* Vital signs - every visit, pre- and post-challenge
* Physical examination - at Screening and Follow up
* Objective ocular measurements performed in the following order so that one does not affect the other:

  * Break up time (BUT): Tear break up time will be measured following the guidelines published in the Report of the International Dry Eye Work Shop (DEWS) 2007.13
  * Staining of the conjunctiva with lissamine green: it stains epithelial cells only if the cell membrane is damaged.
  * Staining of the cornea with fluorescein: Principally for assessing corneal damage, fluorescein should be instilled in a similar way, but with the excess saline on the strip shaken off to instill a minimal volume.
  * Conjunctival chemosis: Lid-parallel conjunctival folds (LIPCOF) will be evaluated with a slit-lamp microscope.
  * Conjunctival redness: The most common clinical sign that is suggestive of ocular surface inflammation is conjunctival redness. Ocular redness can be easily detected with a pen torch or standard slit lamp biomicroscopic examination.
  * Slit lamp microscopy: Assessment of eyelid edema and conjunctival papillae.
  * Assessment of intraocular pressure (IOP) measured with tonometer.
  * Assessment of further ocular symptoms including itching, blurred vision, grittiness.
* Safety laboratory assessments: Complete blood count with differential, blood chemistry, liver function, urine dipstick test - at screening visit, serology at screening and drug of abuse test on investigator's decision
* Skin Prick Test with skin prick test solution (Manufacturer Allergopharma) - at Screening or within the previous 12 months
* Specific CAP analysis (g6) - at Screening or within the previous 12 months
* Vital signs, physical examination and ECG - at screening and follow-up visit
* Adverse events - throughout the study
* Concomitant medication - throughout the study

One to two weeks after the final provocation session, subjects will complete the trial after their follow up visit.

The trial design is appropriate for the indication studied. Validated methods of data collection, analysis, and evaluation will be used for the trial.

The trial endpoints are listed below:

Primary efficacy endpoint:

The primary efficacy endpoint will be the mean 'Total Ocular Symptom Score' (TOSS), calculated as the baseline adjusted mean of TOSS measured every 15 minutes during the grass pollen allergen exposure challenge from time-point 0 to 4 hours on day 8.

TOSS is defined as the sum of the four individual ocular symptoms:

* ocular redness
* ocular itching
* watery eye
* gritty feeling

each scored on a 4-point categorical scale from 0-3 with

"0"= none "1"=mild "2"=moderate "3"=severe

Secondary efficacy endpoints:

* Change in ocular redness image score
* Total nasal symptom score (TNSS) is the sum of the symptoms "nasal congestion", "rhinorrhea"", "itchy nose" and "sneezing".
* Total respiratory symptom score (TRSS) is the sum of the symptoms "cough", "wheeze", "dyspnea".
* Nasal airflow (AAR) will be assessed every 60 minutes during the four hours grass pollen allergen exposure challenge

Each individual symptom of TNSS and TRSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none, "1"=mild, "2"=moderate, "3"=severe). TNSS and TRSS will be assessed every 15 minutes during the four hours grass pollen allergen exposure challenge.

Safety endpoints:

* Adverse events (AEs)
* Safety laboratory
* ECG
* Spirometry (FeV1, FVC)
* Ocular assessments

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Written informed consent obtained before any trial related procedures are performed
* Healthy male or female subjects aged 18 to 65 years
* Female subjects of child-bearing potential must have a negative pregnancy test and be willing to practice appropriate and safe contraceptive methods until the end of treatment visit
* A documented clinically relevant allergic history of moderate to severe SAR with rhinoconjunctivitis to grass pollen for the previous two years
* Subjects exhibit a moderate to severe response to approximately 1800 grass pollen grains/m3 within the first 2 hours in the Vienna Challenge Chamber, which is defined as total ocular symptom score (TOSS) of at least 4 (out of 12) with at least one single ocular symptom scored ≥2 ("moderate") at least twice during the first two hours of the screening challenge session using standard VCC grass pollen allergen mixture. Ocular symptom score is the sum of "ocular redness", "ocular itching", "watery eyes", "gritty feeling" each of which have been scored on a categorical scale from 0 to 3.
* Positive Skin Prick Test (SPT) response (wheal diameter at least 3 mm larger than diluent control) to grass pollen SPT solutions (standard Allergopharma) at screening or within the last 12 months prior to study start.
* Positive serum specific IgE against recombinant major allergen components of the used grass pollen e.g. g6 (specific CAP IgE ≥0.70 kU/L) at screening or within the last 12 months prior to study start.
* Non-smoking subjects (smoked <10 packs per year in their lifetime and had not smoked in the last 6 months).
* Asthma patients only if the asthma condition is mild or intermittent, and if those are not treated with steroids
* Subject has a forced expiratory volume in 1 second (FEV1) of at least 80% of predicted value (ECCS) at the screening.
* Subject is capable of understanding the study procedures and potential risks associated with the study, and voluntarily agrees to participate by giving written informed consent.
* Subject is able to adhere to dose and visit schedules.
* Subject is able to read, understand and complete questionnaires and diaries.

Exclusion Criteria:

A subject meeting any of the exclusion criteria listed below must be excluded from participating in the trial:

* Pregnant, lactating or sexually active women with childbearing potential who are not using a medically accepted and safe birth control method (pregnancy to be controlled by a pregnancy dipstick test).
* Contact lens users
* A clinical history of uncontrolled asthma within 3 months prior to screening.
* Subjects with asthma requiring treatment with inhaled or oral corticosteroids on a regular basis judged by the investigator
* Previous successful immunotherapy to grass pollen, a grass pollen allergen or a cross-reacting allergen within the past 3 years
* Ongoing treatment with any allergen-specific immunotherapy product
* Subjects with a current oral candidiasis infection or treatment for oral candidiasis during the last 30 days before starting the study.
* Subjects with history of tuberculosis.
* Subjects with any fungal/viral/bacterial respiratory or systemic infections during the last 30 days.
* Symptoms of or treatment for upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process (at randomization)
* Subjects with uveitis, prior chemical burn to the ocular surface, pemphigoid, Mooren's ulcer, ulcerative keratitis, bacterial/fungal/viral infection of the eye
* Subjects using any ophthalmic steroids during the last 30 days
* Subjects treated with nasal, inhaled or systemic immunosuppressants during the last 30 days
* History of anaphylaxis with cardiorespiratory symptoms (immunotherapy, exercise induced, food allergy, drugs or an idiopathic reaction).
* Any clinically relevant chronic disease judged by the investigator.
* Systemic or ocular disease involving the immune system judged by the investigator.
* Use of an investigational drug within 30 days/5 half-lives of the drug (which ever longest) prior to screening.
* History of allergy, hypersensitivity or intolerance to any ingredients of the IMP.
* History of alcohol or drug abuse
* Being immediate family of the investigator or trial staff, defined as the investigator's/staff's spouse, parent, child, grandparent or grandchild.
* Subjects treated with topical anti-allergy or cyclosporin-containing eyedrops within 2 weeks before study start
* Subjects treated with leukotriene antagonists (1 month before study start), long- lasting anti-histamines, like cetirizine, fexofenadine, loratadine, desloratadine, hydroxyzine (5 to 10 days before study start), mast cell stabilizer (2 weeks before study start) or nasal decongestant (3 days before study start)
* Subjects with hypersensitivity to immunosuppressants judged by the investigator.
* Presence or history of any ocular infection or clinically significant inflammation
* Ocular surgery in the 3 months preceding the study
* Treatment with corticosteroids in the 4 weeks preceding the study
* Is currently being treated with a medication that induces or inhibits CYP3A4 or 5

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2020-08-04 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Total Ocular Symptom Score | 0-4 hours of allergen challenge
  The total ocular symptom score is the sum of four eye symptoms 'red eyes', 'itchy eyes', and 'watery eyes' and 'gritty feeling' scored every 15 minutes on a categorical scale from 0 (none) to 3 (severe) on challenge day at the times described in the Time and Events Schedule

SECONDARY OUTCOMES:
Total nasal symptom score (TNSS) | 0-4 hours of allergen challenge
  Total nasal symptom score (TNSS) is the sum of the symptoms "nasal congestion", "rhinorrhea"", "itchy nose" and "sneezing".
  Each individual symptom of TNSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none, "1"=mild, "2"=moderate, "3"=severe). TNSS will be assessed every 15 minutes during the four hours grass pollen allergen exposure challenge.
Total respiratory symptom score (TRSS) | 0-4 hours of allergen challenge
  Total respiratory symptom score (TRSS) is the sum of the symptoms "cough", "wheeze", "dyspnea".
  Each individual symptom of TRSS will be scored on a 4-point categorical scale from 0-3 (where "0"= none, "1"=mild, "2"=moderate, "3"=severe). TRSS will be assessed every 15 minutes during the four hours grass pollen allergen exposure challenge.
Nasal airflow (AAR) | 0-4 hours of allergen challenge
  Nasal airflow (AAR) will be assessed every 60 minutes during the four hours grass pollen allergen exposure challenge
change in ocular redness image score | 0-4 hours of allergen challenge
  change in ocular redness image score

CONTACTS AND LOCATIONS:
Overall Officials: Eva Prieschl-Grassauer, PhD, Study Chair — CSO
Locations (1):
- Vienna Challenge Chamber, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sladek S, Unger-Manhart N, Siegl C, Dellago H, Zieglmayer PU, Lemell P, Savli M, Zieglmayer R, Geitzenauer W, Langauer M, Prieschl-Grassauer E. Alleviation of Allergic Rhinoconjunctivitis Symptoms in Participants Treated with a 0.005% Tacrolimus Eye-Drop Solution. Clin Ophthalmol. 2024 Oct 5;18:2797-2811. doi: 10.2147/OPTH.S476163. eCollection 2024. PMID 39386177